CLINICAL TRIAL: NCT06941051
Title: Evaluation of Food Sustainability Knowledge and Attitudes Toward the EAT-Lancet Dietary Pattern Among Turkish Adults
Brief Title: Food Sustainability Knowledge and EAT-Lancet Adherence in Turkish Adults
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL008
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Health Adults
Keywords: Sustainable nutrition; EAT-Lancet; Food sustainability knowledge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health adults: Group/Cohort Description: The study included 3446 individuals aged 19-65. Data were collected using a demographic survey and Food Sustainability Knowledge and Attitudes Questionnaire. Food Consumption Frequency was used to calculate the EAT lancet index.

SUMMARY:
This study aimed to evaluate the knowledge and attitudes of Turkish adults toward food sustainability and assess their adherence to the EAT-Lancet dietary pattern. A cross-sectional study was conducted among 3,446 adults aged 19-65 in Türkiye. Data were collected using a demographic questionnaire, the Food Sustainability Knowledge and Attitudes Questionnaire (FSKAQ), and a food frequency questionnaire to calculate EAT-Lancet index scores. Statistical analyses included Kruskal-Wallis tests, chi-square tests, and multinomial logistic regression.

DETAILED DESCRIPTION:
Objective:

This study aimed to evaluate the knowledge and attitudes of Turkish adults regarding food sustainability and to assess their level of adherence to the EAT-Lancet dietary pattern, a model developed to promote both human health and environmental sustainability.

Methods:

A descriptive, cross-sectional study was conducted across Türkiye with a sample of 3,446 individuals aged between 19 and 65 years. Participants were recruited through voluntary participation, and individuals with chronic illnesses, alcohol or substance dependency, or illiteracy were excluded. Data were collected using a structured questionnaire that included demographic variables (e.g., age, gender, marital status, income, physical activity), anthropometric measurements (height and weight), and dietary intake.

Participants' knowledge and attitudes toward food sustainability were assessed using the Food Sustainability Knowledge and Attitudes Questionnaire (FSKAQ), which has been validated in Turkish. This instrument consists of four sub-dimensions addressing different aspects of sustainability knowledge and attitudes but does not yield a total score. Each sub-dimension is evaluated individually.

Dietary intake was assessed using a food frequency questionnaire (FFQ), and adherence to the EAT-Lancet dietary pattern was calculated using the EAT-Lancet index. This index includes 14 food components categorized as "emphasized" or "restricted" foods and assigns scores from 0 to 3 for each, with higher total scores indicating greater adherence. Final scores were divided into quartiles (Q1-Q4) to classify adherence levels.

All statistical analyses were conducted using SPSS 26.0. Descriptive statistics were used to summarize participant characteristics. The Kruskal-Wallis H test and chi-square tests were used for group comparisons, and multinomial logistic regression was applied to identify factors associated with higher EAT-Lancet index adherence. A significance level of p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals residing in Türkiye,
* Aged between 19 and 64 years,
* Voluntarily agreed to participate in the study,
* Completed the questionnaire in full,
* Provided complete anthropometric, demographic, and dietary data.

Exclusion Criteria:

* Individuals with alcohol or substance dependence,
* Those diagnosed with chronic diseases (e.g., diabetes, hypertension, cardiovascular disease),
* Illiterate individuals,
* Participants with incomplete questionnaire responses or missing anthropometric or dietary data.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample in Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 3446 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Food Sustainability Knowledge and Attitudes Questionnaire | Baseline
  This scale was designed to assess participants' knowledge and attitudes toward sustainable nutrition and consists of a total of 7 questions (5 related to knowledge and 2 to attitudes). The scale includes four sub-dimensions: Knowledge of Sustainability and Sustainable Nutrition (9 items), Knowledge of Statements Defining a Sustainable Diet (12 items), Knowledge of Planetary Health and Sustainability (10 items), and Attitudes Toward Sustainable Nutrition (2 items). The scale does not yield a total score; only specific sub-dimensions are scored independently. The "Knowledge of Statements Defining a Sustainable Diet" sub-dimension, designed in Likert type, is scored item by item. In the "Knowledge of Planetary Health and Sustainability" dimension, only the second section is scored. In the "Attitudes Toward Sustainable Nutrition" sub-dimension, each of the two items is scored separately. The remaining questions are not scored.
EAT-Lancet Index | Baseline
  EAT-Lancet Index:
  The EAT-Lancet Index evaluates adherence to a sustainable and healthy diet through 14 food components, categorized as either "restricted" (e.g., red meat, poultry, eggs, added sugars) or "emphasized" (e.g., fruits, vegetables, legumes, whole grains, nuts, fish). Intakes are assessed in grams per day (uncooked weight). Each component is scored from 0 (low adherence) to 3 (high adherence), with a total possible score ranging from 0 to 42. Scores were divided into quartiles (Q1-Q4) to indicate adherence levels. Food frequency questionnaire data were used for calculation.

SECONDARY OUTCOMES:
Food Consumption Frequency | Baseline
  It was used to determine how often and how much of food groups or nutrients were consumed. Consumption frequency was given as day, month or week. Food groups include milk and dairy products, meat-egg-legumes, vegetables and fruits, grains and oilseeds. Participants were asked how often they consumed which food (everyday, 5-6 times a week, 3-4 times a week, 1-2 times a week, 1 time in 15 days, 1 time in a month, 1 time in 3 months, 1 time in 6 months, never) and used for EAT lancet index calculation.
Sociodemographic characteristics | Baseline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No